CLINICAL TRIAL: NCT00898963
Title: Identification of Biomarkers in Follicular Lymphoma
Brief Title: Biomarkers in Patients With Stage III or Stage IV Follicular Lymphoma Treated on Clinical Trial E-1496
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000544400; ECOG-E1496T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Gene Expression Profiling; Microarray Analysis; Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry; Immunologic Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: polymorphism analysis
Other: diagnostic laboratory biomarker analysis
Other: immunohistochemistry staining method
Other: immunologic technique

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how patients respond to treatment.

PURPOSE: This laboratory study is looking at biomarkers in patients with stage III or stage IV follicular lymphoma treated on clinical trial E-1496.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate gene expression profiles with progression-free survival (PFS) of patients with stage III or IV follicular lymphoma treated with cyclophosphamide, vincristine, and prednisone with or without rituximab on clinical trial E-1496.
* Determine if immunoglobulin Fc-gamma receptor polymorphisms are predictive of PFS in these patients.
* Assess the significance of the microenvironment by constructing tissue microarrays of follicular lymphoma and immunostaining with relevant biomarkers.
* Correlate relevant biomarkers with clinical features, response, and PFS.

OUTLINE: This is a multicenter study.

Tissue samples are analyzed by gene expression profiling, microarrays to predict gene expression, immunohistochemistry, and immunoglobulin Fc-gamma receptor polymorphism analysis for biological markers.

PROJECTED ACCRUAL: A total of 175 samples will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of follicular lymphoma

  * Stage III or IV disease
* Received cyclophosphamide, vincristine, and prednisone with or without rituximab on clinical trial E-1496

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E1496
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2007-04-18 (Actual); Primary Completion 2011-02-11 (Actual); Study Completion 2011-02-11 (Actual)

PRIMARY OUTCOMES:
Correlation of gene expression profiles with progression-free survival (PFS) | 1 month
Prediction of PFS by immunoglobulin Fc-gamma receptor polymorphisms as assessed by immunohistochemistry | 1 month
Assessment of significance of microenvironment by constructing tissue microarrays and immunostaining with relevant biomarkers | 1 month
Correlation of relevant biomarkers with clinical features, response, and PFS | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Randall D. Gascoyne, MD, Study Chair — British Columbia Cancer Agency